CLINICAL TRIAL: NCT01468922
Title: Phase Ib Study of the Combination of Pazopanib, an Oral VEGFR Inhibitor, and ARQ 197 (Tivantinib), an Oral MET Inhibitor, in Patients With Refractory Advanced Solid Tumors
Brief Title: Pazopanib and ARQ 197 for Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Alice Chen, M.D., Principal Investigator, National Cancer Institute (NCI)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 120009; 12-C-0009
Record Dates: First submitted 2011-11-08; First posted 2011-11-10 (Estimated); Results first posted 2022-07-01 (Actual); Last update posted 2022-07-01 (Actual); Status verified 2022-06

CONDITIONS: Solid Tumor
Keywords: Pazopanib; Tivantinib; MET Inhibitor; Advanced Cancer; Anti-Angiogenesis; Cancer; Solid Tumor; Sarcoma
MeSH Terms: conditions — Neoplasms; Sarcoma | interventions — pazopanib; ARQ 197

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- A/Combination pazopanib plus ARQ 197 (Tivantinib) (Experimental): Combination pazopanib plus ARQ197 at doses established during escalation phase
  Interventions: Drug: Pazopanib; Drug: ARQ 197

INTERVENTIONS:
Drug: Pazopanib — Vascular endothelial growth factor (VEGFR) inhibitor
  Other Names: Votrient
Drug: ARQ 197 — Hepatocyte growth factor receptor (mesenchymal-epithelial transition factor [c-MET]) inhibitor
  Other Names: Tivantinib

SUMMARY:
Background:

- Pazopanib is an anticancer drug that blocks the growth of new blood vessels in tumors. It has been approved to treat renal cell cancer and soft tissue sarcomas in patients who have received prior chemotherapy. ARQ 197 (Tivantinib) is an experimental drug that blocks a protein called mesenchymal-epithelial transition factor (c-MET), which cancer cells need to grow. Studies suggest that some drugs that block blood vessel growth can increase the production of c-MET in tumors, which helps cancer cells keep growing. Blocking both blood vessel growth and c-MET with pazopanib and ARQ 197 may help kill cancer cells faster. This study will use these drugs to treat solid tumors that have not responded to earlier treatments.

Objectives:

- To test the safety and effectiveness of pazopanib and ARQ 197 for advanced solid tumors.

Eligibility:

- Individuals at least 18 years of age who have advanced solid tumors that have not responded to earlier treatments.

Design:

* Participants will be screened with a physical exam and medical history. They will also have blood and urine tests, and imaging studies.
* The study drugs will be given in 4-week cycles of treatment. Participants will take pazopanib once a day and ARQ 197 twice a day by mouth. Some participants will start with pazopanib or ARQ 197 alone for the first week. Then they will take both drugs together for the rest of the study.
* Participants will be monitored with frequent blood tests and imaging studies. Optional tumor samples may be collected during different treatment cycles.

DETAILED DESCRIPTION:
Background:

* Vascular endothelial growth factor (VEGF) and hepatocyte growth factor (HGF) signal transduction pathways have synergistic effects on promoting angiogenesis and growth factor expression. Hypoxia caused by treatment with VEGF inhibitors results in the upregulation of mesenchymal-epithelial transition factor (c-MET), the receptor for HGF. In a mouse model, combined blockade of VEGFR and c-MET significantly prolonged survival compared with inhibition of either target alone.
* We hypothesize that co-administration of the putative hepatocyte growth factor receptor (MET) inhibitor ARQ 197 (Tivantinib) will prevent the adaptive response to hypoxia resulting from treatment with the VEGFR inhibitor pazopanib, and conversely, that co-administration of pazopanib will prevent the effect of increased VEGF and reduced thrombospondin 1 in tumors after treatment with ARQ 197. Therefore, the combination of these agents may result in improved antitumor effects.

Objectives:

* Establish the safety and tolerability of the combination of pazopanib with ARQ 197 in patients with refractory advanced solid tumors.
* Establish the maximum tolerated dose (MTD) of the combination of pazopanib with ARQ 197 in patients with refractory advanced solid tumors.
* Evaluate changes in MET and phospho-MET following treatment with pazopanib and ARQ 197 in patients with refractory advanced solid tumors.
* Determine the pharmacokinetics (PK) of pazopanib and ARQ 197.
* Determine and compare levels of total MET, phospho MET, Hypoxia-Inducible Factor (HIF)-1, and epithelial-mesenchymal transition markers (e-cadherin, beta catenin) in tumor biopsy samples prior to and following administration of the study drugs.
* Determine and compare levels of circulating levels of hepatocyte growth factor (HGF), soluble MET (sMET), vascular endothelial growth factor A (VEGF-A), and soluble vascular endothelial growth factor receptor 2 (VEGFR2) (sVEGFR2) prior to and following administration of the study drugs.
* Determine polymorphisms in the cytochrome P450 2C19 (CYP2C19) and correlate these with the observed toxicities, and the pharmacokinetics (PK) of ARQ 197.
* Evaluate antitumor activity of the combination of pazopanib and ARQ 197 in patients with refractory advanced solid tumors.

Eligibility:

-Adults with advanced, refractory solid tumors. Patients enrolling in the expansion cohorts must have advanced sarcoma, gastric cancer, and MET-expressing malignancies, have disease amenable to biopsy, and be willing to undergo pre-and post-treatment biopsies.

Study Design:

* ARQ 197 will be administered orally twice daily and pazopanib orally once daily, in 28-day cycles.
* Dose escalation will proceed using the traditional 3+3 design.
* Once the maximum tolerated dose (MTD) is established, an additional cohort will be accrued for pharmacodynamic (PD) studies in tumor biopsies (required in the expansion phase). For the first week, patients will receive pazopanib alone to compare PK and PD results; combination therapy will be given from week 2 onwards.

ELIGIBILITY:
* ELIGIBILITY CRITERIA:
* Patients with histologically confirmed (by the Laboratory of Pathology, National Institutes of Health (NIH) solid tumors that have progressed following at least one line of standard therapy or for whom no standard treatment options exist.
* Patients must have measurable or evaluable disease.
* Patients enrolling in the expansion cohorts must have disease amenable to biopsy, and be willing to undergo pre-and post-treatment biopsies.
* Patients must have completed any chemotherapy, radiation therapy, or biologic therapy greater than or equal to 4 weeks prior to entering the study (6 weeks for nitrosoureas or mitomycin C). Patients must be greater than or equal to 2 weeks since any prior administration of a study drug in a phase 0 or equivalent study. Patients must have recovered to eligibility levels from prior toxicity or adverse events. Treatment with bisphosphonates is permitted.
* Patients who have had prior treatment with any anti-angiogenic therapy and/or mesenchymal epithelial transition factor (c-MET) inhibitor are eligible in the dose escalation phase unless the antiangiogenic therapy and/or c-MET inhibitor were administered within the 4 weeks prior to entering the study. In the expansion phase, prior c-MET inhibitor is not allowed, and anti-angiogenic therapy is allowed unless it was administered within the 3 months prior to entering the study.
* Age greater than or equal to 18 years. Because no dosing or adverse event data are currently available on the use of pazopanib in combination with ARQ 197 (Tivantinib) in patients less than 18 years of age, children are excluded from this study.
* Life expectancy greater than 3 months.
* Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1.
* Patients must have normal organ and marrow function as defined below:

  * Absolute neutrophil count greater than or equal to 1,500/microL
  * Platelets greater than or equal to 100,000/microL
  * Total bilirubin less than or equal to 1.5 X institutional upper limit of normal (ULN)
  * Aspartate aminotransferase (AST) serum glutamic oxaloacetic transaminase(SGOT)/alanine transaminase (ALT) serum glutamic pyruvic transaminase(SGPT) less than or equal to 2.5 X institutional ULN
  * Creatinine less than or equal to 1.5 mg/dL (133 mcmol/L); OR
  * Measured creatinine greater than or equal to 60 mL/minute for patients with clearance creatinine levels greater than 1.5 mg/dL
  * Urine protein/creatinine ratio less than 1 OR 24-hour urine protein less than 1 gram
* Subjects who have both bilirubin greater than ULN and AST/ALT greater than ULN are not eligible.
* Subjects in the expansion cohort must have prothrombin time (PT)/ international normalized ratio (INR)/partial thromboplastin time (PTT) less than or equal to 1.2 X institutional ULN, except patients with confirmed positive lupus anticoagulant test.
* Subjects must have blood pressure (BP) no greater than 140 mmHg (systolic) and 90 mmHg (diastolic) for eligibility. Initiation or adjustment of BP medication is permitted prior to study entry provided that the average of three BP readings at a visit prior to enrollment is less than 140/90 mmHg.
* The effects of study drugs on the developing human fetus are unknown. For this reason, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study participation, and for at least 2 months after dosing with study drugs ceases. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately. Women of child-bearing potential must have a negative pregnancy test prior to entry.
* Patients must be able to swallow whole tablets or capsules. Nasogastric or G-tube administration is not allowed.
* Ability to understand and the willingness to sign a written informed consent document.

EXCLUSION CRITERIA:

* Patients who are receiving any other investigational agents.
* Patients with active brain metastases or carcinomatous meningitis are excluded from this clinical trial. Patients whose brain metastatic disease status has remained stable for greater than or equal to 4 weeks following treatment of the brain metastases are eligible to participate.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to pazopanib or ARQ 197.
* Eligibility of subjects receiving any medications or substances known to affect or with the potential to affect the activity or pharmacokinetics of pazopanib or ARQ 197 will be determined following review of their cases by the Principal Investigator. Efforts should be made to switch subjects with gliomas or brain metastases who are taking enzyme inducing anticonvulsant agents to other medications.
* Certain medications that act through the cytochromes P450 (CYP450) system are specifically prohibited in subjects receiving pazopanib and ARQ 197 and others should be avoided or administered with extreme caution.

  * Strong inhibitors of cytochrome P450 3A4 (CYP3A4) such as ketoconazole, itraconazole, clarithromycin, atazanavir, indinavir, nefazodone, nelfinavir, ritonavir, saquinavir, telithromycin, voriconazole may increase pazopanib concentrations and are prohibited; although, in exceptional circumstances they may be administered in conjunction with lowering the dose of pazopanib by 50% of what would otherwise be administered. Grapefruit juice is also an inhibitor of CYP450 and should not be taken with pazopanib.
  * Strong inducers of Cytochrome P450 Family 3 Subfamily A Member 4 (CYP3A4), such as rifampin, may decrease pazopanib concentrations, are strictly prohibited.
  * Medications which have narrow therapeutic windows and are substrates of CYP3A4, cytochrome P450 2D6 CYP2D6), or cytochrome P₄₅₀2C8 (CYP2C8) should be avoided and, if necessary, administered with caution.
  * Inhibitors or inducers of cytochrome P450 2C19 (CYP2C19) should be avoided and, if necessary, administered with caution.
* Cardiovascular baseline corrected QT Interval (QTc) greater than or equal to 480 msec will exclude patients from entry on study. Medications that may cause QTc interval prolongation are listed, and should be avoided by patients entering on trial. Patients for whom a given medication that may cause QTc interval prolongation cannot be discontinued may be eligible at the discretion of the study principal investigator (PI). A comprehensive list of agents with the potential to cause QTc prolongation can be found at http://www.azcert.org/medical-pros/drug-lists/bycategory.cfm. (Note: If subjects must take medications with a risk or possible risk of Torsades de Pointes, they should be watched carefully for symptoms of Torsades de Pointes, such as syncope. Performing additional electrocardiograms (EKGs) on subjects who must take one or more of these medications is not required; however, additional investigations, including EKGs, may be performed as per the treating physicians judgment.)
* Subjects with any of the following cardiovascular conditions within the past 6 months:

  * cerebrovascular accident (CVA) or transient ischemic attack (TIA)
  * clinically significant bradycardia or other uncontrolled cardiac arrhythmia
  * admission for unstable angina or myocardial infarction
  * cardiac angioplasty or stenting
  * coronary artery bypass graft surgery
  * pulmonary embolism, untreated deep venous thrombosis (DVT) or DVT which has been treated with therapeutic anticoagulation for less than 6 weeks
  * arterial thrombosis
  * symptomatic peripheral vascular disease
  * Class III or IV heart failure as defined by the New York Heart Association (NYHA) functional classification system. A subject who has a history of Class II heart failure and is asymptomatic on treatment may be considered eligible

    * History of serious or non-healing wound, ulcer, or bone fracture.
    * Patients who received major surgery within the past 4 weeks
    * Subjects with any condition that may impair the ability to swallow or absorb oral medications/investigational product including:
  * any lesion, whether induced by tumor, radiation or other conditions, which makes it difficult to swallow capsules or pills
  * prior surgical procedures affecting absorption including, but not limited to major resection of stomach or small bowel
  * active peptic ulcer disease
  * malabsorption syndrome
* Subjects with any condition that may increase the risk of gastrointestinal bleeding or gastrointestinal perforation, including

  * active peptic ulcer disease
  * known intraluminal metastatic lesions
  * inflammatory bowel disease (e.g., ulcerative colitis, Crohn's disease) or other gastrointestinal conditions which increase the risk of perforation
  * history of abdominal fistula, gastrointestinal perforation or intraabdominal abscess within 28 days prior to beginning study treatment

    * History of hemoptysis in excess of 2.5 mL (1/2 teaspoon ) within 8 weeks prior to first dose of study drug.
    * Urine protein/creatinine ratio should be screened by urine analysis. If protein is 1+ or higher, 24-hour urine protein should be obtained and the level should be less than 1g for patient enrollment. Patients with less than 1+ proteinuria are eligible following initial determination by urinalysis within 1 week prior to enrollment and do not need the urinalysis repeated.
    * Patients with clinically significant intercurrent illnesses, including but not limited to, life threatening infection, psychiatric illness/social situations that would limit compliance with study requirements will not be eligible to participate.
    * Pregnant women are excluded from this study because the effects of the study drugs on the developing fetus are unknown. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with the study drugs, breastfeeding should be discontinued prior to the first dose of study drug and women should refrain from nursing throughout the treatment period and for 14 days following the last dose of study drug.
    * Human immunodeficiency virus (HIV)-positive patients on combination antiretroviral therapy are ineligible because of the potential for pharmacokinetic (PK) interactions.
    * Patients who require use of coumarin-derivative anticoagulants such as warfarin are excluded. Low molecular weight heparin is permitted for prophylactic use, but not therapeutic use.

INCLUSION OF WOMEN AND MINORITIES:

Both men and women of all races and ethnic groups are eligible for this trial.

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2012-01-23 (Actual); Primary Completion 2014-09-30 (Actual); Study Completion 2016-02-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alice P Chen, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gerritsen ME, Tomlinson JE, Zlot C, Ziman M, Hwang S. Using gene expression profiling to identify the molecular basis of the synergistic actions of hepatocyte growth factor and vascular endothelial growth factor in human endothelial cells. Br J Pharmacol. 2003 Oct;140(4):595-610. doi: 10.1038/sj.bjp.0705494. Epub 2003 Sep 22. PMID 14504135
- [Background] Xin X, Yang S, Ingle G, Zlot C, Rangell L, Kowalski J, Schwall R, Ferrara N, Gerritsen ME. Hepatocyte growth factor enhances vascular endothelial growth factor-induced angiogenesis in vitro and in vivo. Am J Pathol. 2001 Mar;158(3):1111-20. doi: 10.1016/S0002-9440(10)64058-8. PMID 11238059
- [Background] Van Belle E, Witzenbichler B, Chen D, Silver M, Chang L, Schwall R, Isner JM. Potentiated angiogenic effect of scatter factor/hepatocyte growth factor via induction of vascular endothelial growth factor: the case for paracrine amplification of angiogenesis. Circulation. 1998 Feb 3;97(4):381-90. doi: 10.1161/01.cir.97.4.381. PMID 9468212
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2012-C-0009.html

RESULTS

PARTICIPANT FLOW:
Groups:
- Dose Level (DL) 1: Pazopanib (Paz): 400 mg & ARQ 197 (Tivantinib): 120 mg: Cycle=28 days,Pazopanib: 400 mg by mouth (PO) every day (QD) ,ARQ 197: 120 mg PO twice a day (BID)
- Dose Level 2: Pazopanib: 600 mg & ARQ 197: 120 mg: Cycle=28 days,Pazopanib: 600 mg by mouth (PO) every day (QD),ARQ 197: 120 mg by mouth (PO) twice a day (BID)
- Dose Level 3: Pazopanib: 600 mg & ARQ 197: 240 mg: Cycle=28 days,Pazopanib: 600 mg by mouth (PO) every day (QD),ARQ 197: 240 mg by mouth (PO) twice a day (BID)
- DL 3 Followed by DL 2: Pazopanib: 600 mg & ARQ 197: 240 mg Foll/by Pazopanib: 600 mg/ARQ 197:120 mg: Cycle=28 days,Pazopanib: 600 mg by mouth (PO) every day (QD),ARQ 197: 240 mg by mouth (PO) twice a day (BID) foll/by Cycle=28 days,Pazopanib: 600 mg by mouth (PO) every day (QD),ARQ 197: 120 mg by mouth (PO) twice a day (BID)
- Dose Level 4: Pazopanib: 800 mg & ARQ 197: 240 mg: Cycle=28 days,Pazopanib: 800 mg by mouth (PO) every day (QD),ARQ 197: 240 mg by mouth (PO) twice a day (BID)
- DL 4 Followed by DL 3: Pazopanib: 800 mg & ARQ 197: 240 mg Foll/by Pazopanib: 600 mg/ARQ 197: 240 mg: Cycle=28 days,Pazopanib: 800 mg by mouth (PO) every day (QD),ARQ 197: 240 mg by mouth (PO) twice a day (BID) foll/by Cycle=28 days,Pazopanib: 600 mg by mouth (PO) every day (QD),ARQ 197: 240 mg by mouth (PO) twice a day (BID)
- DL4 Foll/by DL3 Foll/by DL2 Paz800mg/ARQ240mg Foll/by Paz600 mg/ARQ240mg Foll/by Paz600 mg/ARQ120 mg: Cycle=28 days,Pazopanib: 800 mg by mouth (PO) every day (QD),ARQ 197: 240 mg by mouth (PO) twice a day (BID) foll/by Cycle=28 days,Pazopanib: 600 mg by mouth (PO) every day (QD),ARQ 197: 240 mg by mouth (PO) twice a day (BID) foll/by Cycle=28 days,Pazopanib: 600 mg by mouth (PO) every day (QD),ARQ 197: 120 mg by mouth (PO) twice a day (BID)
- Dose Level 5: Pazopanib: 800 mg & ARQ 197: 360 mg: Cycle=28 days,Pazopanib: 800 mg by mouth (PO) every day (QD),ARQ 197: 360 mg by mouth (PO) twice a day (BID)
- Enrolled But Not Treated: Enrolled but failed screening and was not treated.
Period: Overall Study
Arm/Group | Dose Level (DL) 1: Pazopanib (Paz): 400 mg & ARQ 197 (Tivantinib): 120 mg | Dose Level 2: Pazopanib: 600 mg & ARQ 197: 120 mg | Dose Level 3: Pazopanib: 600 mg & ARQ 197: 240 mg | DL 3 Followed by DL 2: Pazopanib: 600 mg & ARQ 197: 240 mg Foll/by Pazopanib: 600 mg/ARQ 197:120 mg | Dose Level 4: Pazopanib: 800 mg & ARQ 197: 240 mg | DL 4 Followed by DL 3: Pazopanib: 800 mg & ARQ 197: 240 mg Foll/by Pazopanib: 600 mg/ARQ 197: 240 mg | DL4 Foll/by DL3 Foll/by DL2 Paz800mg/ARQ240mg Foll/by Paz600 mg/ARQ240mg Foll/by Paz600 mg/ARQ120 mg | Dose Level 5: Pazopanib: 800 mg & ARQ 197: 360 mg | Enrolled But Not Treated
Started | 3 | 3 | 2 | 1 | 4 | 1 | 1 | 16 | 1
Completed | 1 | 3 | 2 | 1 | 2 | 1 | 1 | 12 | 0
Not Completed | 2 | 0 | 0 | 0 | 2 | 0 | 0 | 4 | 1
Not completed — Screening failure | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Per patient choice | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Switched to alternative treatment | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Enrolled on new protocol | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Infection of blood | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Patient choice - surgery | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Refused further treatment | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Dose Level (DL) 1: Pazopanib (Paz): 400 mg & ARQ 197: 120 mg: Cycle=28 days,Pazopanib: 400 mg by mouth (PO) every day (QD) ,ARQ 197: 120 mg PO twice a day (BID)
- Total: Total of all reporting groups
Arm/Group | Dose Level (DL) 1: Pazopanib (Paz): 400 mg & ARQ 197: 120 mg | Dose Level 2: Pazopanib: 600 mg & ARQ 197: 120 mg | Dose Level 3: Pazopanib: 600 mg & ARQ 197: 240 mg | DL 3 Followed by DL 2: Pazopanib: 600 mg & ARQ 197: 240 mg Foll/by Pazopanib: 600 mg/ARQ 197:120 mg | Dose Level 4: Pazopanib: 800 mg & ARQ 197: 240 mg | DL 4 Followed by DL 3: Pazopanib: 800 mg & ARQ 197: 240 mg Foll/by Pazopanib: 600 mg/ARQ 197: 240 mg | DL4 Foll/by DL3 Foll/by DL2 Paz800mg/ARQ240mg Foll/by Paz600 mg/ARQ240mg Foll/by Paz600 mg/ARQ120 mg | Dose Level 5: Pazopanib: 800 mg & ARQ 197: 360 mg | Enrolled But Not Treated | Total
Number analyzed (Participants) | 3 | 3 | 2 | 1 | 4 | 1 | 1 | 16 | 1 | 32
Age, Categorical [Count of Participants; unit: Participants] — The collected baseline data for one participant who failed screening is shown here.
  Participants
    <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Between 18 and 65 years | 2 | 3 | 1 | 1 | 4 | 1 | 1 | 15 | 1 | 29
    >=65 years | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 3
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.7 (23.95) | 50.9 (11.92) | 60.3 (7.21) | 27.6 (0) | 56.38 (8.42) | 20.5 (0) | 61.9 (0) | 50.04 (13.45) | 44.4 (0) | 49.25 (14.56)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 1 | 0 | 1 | 1 | 0 | 9 | 1 | 14
  Male | 3 | 2 | 1 | 1 | 3 | 0 | 1 | 7 | 0 | 18
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 2 | 0 | 4
  Not Hispanic or Latino | 3 | 3 | 2 | 0 | 4 | 0 | 1 | 14 | 1 | 28
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Asian | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 3 | 0 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 3
  White | 3 | 3 | 1 | 0 | 3 | 1 | 0 | 8 | 1 | 20
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 3
Region of Enrollment [Number; unit: participants]
  United States | 3 | 3 | 2 | 1 | 4 | 1 | 1 | 16 | 1 | 32

OUTCOME MEASURES:

1. Primary Outcome: Number of Grade 3 or 4 Adverse Events, Highest Occurrence Per Participant
Description: The highest Grade 3 or 4 adverse events were assessed by the Common Terminology Criteria for Adverse Events (CTCAE v4.0). Grade 3 is severe, and Grade 4 is life threatening.
Time Frame: Time receiving study drug, up to 22 cycles
Measure: Number; unit: Adverse events
Arm/Group | Dose Level (DL) 1: Pazopanib (Paz): 400 mg & ARQ 197: 120 mg | Dose Level 2: Pazopanib: 600 mg & ARQ 197: 120 mg | Dose Level 3: Pazopanib: 600 mg & ARQ 197: 240 mg | DL 3 Followed by DL 2: Pazopanib: 600 mg & ARQ 197: 240 mg Foll/by Pazopanib: 600 mg/ARQ 197:120 mg | Dose Level 4: Pazopanib: 800 mg & ARQ 197: 240 mg | DL 4 Followed by DL 3: Pazopanib: 800 mg & ARQ 197: 240 mg Foll/by Pazopanib: 600 mg/ARQ 197: 240 mg | DL4 Foll/by DL3 Foll/by DL2 Paz800mg/ARQ240mg Foll/by Paz600 mg/ARQ240mg Foll/by Paz600 mg/ARQ120 mg | Dose Level 5: Pazopanib: 800 mg & ARQ 197: 360 mg
Number analyzed (Participants) | 3 | 3 | 2 | 1 | 4 | 1 | 1 | 16
Adverse events
  Grade 3 | 1 | 0 | 0 | 0 | 3 | 5 | 1 | 7
  Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 10

2. Primary Outcome: Changes in MET and Phospho-MET Levels
Description: MET or phospho-MET levels (in fmol) normalized to the amount of total protein in a sample (in mg).
Time Frame: MET and phospho-MET levels were measured on Cycle 1 Day 1 and Cycle 1 Day 8.
Population: Biopsies were not collected for this assay from all participants, and not all biopsies yielded quantifiable data. While biopsies were collected from 8 patients at Dose Level 5, not every biopsy pair yielded a quantifiable signal in these assays. There were 5 pairs averaged for the intact MET and 2 pairs each for the pY1234/1235-MET and pY1356-MET. Unquantifiable biopsy pairs (either at one or both time points) were excluded from the analysis.
Measure: Mean (Standard Deviation); unit: fmol/mg
Units Other Than Participants: Collected biopsy pairs
Arm/Group | Dose Level (DL) 1: Pazopanib (Paz): 400 mg & ARQ 197: 120 mg | Dose Level 2: Pazopanib: 600 mg & ARQ 197: 120 mg | Dose Level 3: Pazopanib: 600 mg & ARQ 197: 240 mg | DL 3 Followed by DL 2: Pazopanib: 600 mg & ARQ 197: 240 mg Foll/by Pazopanib: 600 mg/ARQ 197:120 mg | Dose Level 4: Pazopanib: 800 mg & ARQ 197: 240 mg | DL 4 Followed by DL 3: Pazopanib: 800 mg & ARQ 197: 240 mg Foll/by Pazopanib: 600 mg/ARQ 197: 240 mg | DL4 Foll/by DL3 Foll/by DL2 Paz800mg/ARQ240mg Foll/by Paz600 mg/ARQ240mg Foll/by Paz600 mg/ARQ120 mg | Dose Level 5: Pazopanib: 800 mg & ARQ 197: 360 mg
Number analyzed (Participants) | 3 | 3 | 2 | 1 | 4 | 1 | 0 | 8
Number analyzed (Collected biopsy pairs) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 8
fmol/mg
  Intact MET: number analyzed (Collected biopsy pairs) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 5
  Intact MET | -52.66 (NA) — Not all biopsies yielded quantifiable data. Standard deviation was not calculated because only 1 biopsy pair was analyzed; calculating standard deviation requires at least 2 measured values. |  |  |  |  |  |  | -195.4 (218.9)
  pY1234/1235-MET: number analyzed (Collected biopsy pairs) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2
  pY1234/1235-MET | NA — Not all biopsies yielded quantifiable data. No biopsy pairs yielded quantifiable data for pY1234/1235-MET. |  |  |  |  |  |  | -130.3 (40.2)
  pY1356-MET: number analyzed (Collected biopsy pairs) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2
  pY1356-MET | NA — Not all biopsies yielded quantifiable data. No biopsy pairs yielded quantifiable data for pY1234/1235-MET. |  |  |  |  |  |  | -51.5 (1.8)

3. Other Pre Specified Outcome: Number of Participants With Serious and Non-serious Adverse Events Assessed by the Common Terminology Criteria for Adverse Events (CTCAE v4.0)
Description: Here is the number of participants with serious and non-serious adverse events assessed by the Common Terminology Criteria for Adverse Events (CTCAE v4.0). A non-serious adverse event is any untoward medical occurrence. A serious adverse event is an adverse event or suspected adverse reaction that results in death, a life-threatening adverse drug experience, hospitalization, disruption of the ability to conduct normal life functions, congenital anomaly/birth defect or important medical events that jeopardize the patient or subject and may require medical or surgical intervention to prevent one of the previous outcomes mentioned.
Time Frame: Date treatment consent signed to date off study, approx 22m (month)/2 days(d); 13m/20 d; 5m/23 d; 17m./24 d; 7 m/5 d; 5m/5 d; 5m/13 d; and 23m/21d for DL1, DL2, DL3, DL3 foll/by DL2, DL4, DL4 foll/by DL3, DL 4 foll/by DL 3 foll/by DL2; & DL5 respectively.
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Level (DL) 1: Pazopanib (Paz): 400 mg & ARQ 197: 120 mg | Dose Level 2: Pazopanib: 600 mg & ARQ 197: 120 mg | Dose Level 3: Pazopanib: 600 mg & ARQ 197: 240 mg | DL 3 Followed by DL 2: Pazopanib: 600 mg & ARQ 197: 240 mg Foll/by Pazopanib: 600 mg/ARQ 197:120 mg | Dose Level 4: Pazopanib: 800 mg & ARQ 197: 240 mg | DL 4 Followed by DL 3: Pazopanib: 800 mg & ARQ 197: 240 mg Foll/by Pazopanib: 600 mg/ARQ 197: 240 mg | DL4 Foll/by DL3 Foll/by DL2 Paz800mg/ARQ240mg Foll/by Paz600 mg/ARQ240mg Foll/by Paz600 mg/ARQ120 mg | Dose Level 5: Pazopanib: 800 mg & ARQ 197: 360 mg
Number analyzed (Participants) | 3 | 3 | 2 | 1 | 4 | 1 | 1 | 16
Participants | 3 | 3 | 2 | 1 | 4 | 1 | 1 | 16

4. Other Pre Specified Outcome: Pazopanib-induced Changes to Epithelial-mesenchymal Phenotype in Human Tumors
Description: Core tumor biopsies were collected from participants with advanced malignancies. Analyses was performed by epithelial-mesenchymal transition immunofluorescence assay (EMT-IFA) for changes in E-cadherin (E+), vimentin(V+), and mixed V+E+ phenotypes. The small imaging pixel size (0.25 µm^2)of the IFA relative to the dimensions of the cross sectional areas of tumor (ranging from 75 to 500 µm^2 in parotid, prostate, colon, and ovarian cancers) allowed us to quantify individual areas of V+ and E+ staining as well as areas of colocalized E+V+ staining within single cells. The assay reports the change in log10(V/E) vratios. The log10(V/E) ratio was determined pre-treatment and in day 8 biopsies and the reported values indicate the change between the two time points. Each value in the table as currently written reflects the change in log10(V/E) ratios between pre- and post-treatment E-cadherin and vimentin values. The full range values indicate the range of changes observed for individual pt.
Time Frame: Pre-treatment and day 8 post administration
Population: This analysis was only performed on biopsy pairs from participants at Dose Level 5, so no biopsy pairs were collected at other Dose Levels (which is why the other levels indicate 0 participants analyzed) and analysis of the changes at those Dose Levels was not applicable (N/A) since no samples were collected.
Measure: Mean (Full Range); unit: Change in log10(V/E) Ratios
Arm/Group | Dose Level (DL) 1: Pazopanib (Paz): 400 mg & ARQ 197: 120 mg | Dose Level 2: Pazopanib: 600 mg & ARQ 197: 120 mg | Dose Level 3: Pazopanib: 600 mg & ARQ 197: 240 mg | DL 3 Followed by DL 2: Pazopanib: 600 mg & ARQ 197: 240 mg Foll/by Pazopanib: 600 mg/ARQ 197:120 mg | Dose Level 4: Pazopanib: 800 mg & ARQ 197: 240 mg | DL 4 Followed by DL 3: Pazopanib: 800 mg & ARQ 197: 240 mg Foll/by Pazopanib: 600 mg/ARQ 197: 240 mg | DL4 Foll/by DL3 Foll/by DL2 Paz800mg/ARQ240mg Foll/by Paz600 mg/ARQ240mg Foll/by Paz600 mg/ARQ120 mg | Dose Level 5: Pazopanib: 800 mg & ARQ 197: 360 mg
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 7
Change in log10(V/E) Ratios |  |  |  |  |  |  |  | 0.332 [-0.126 to 0.723]

ADVERSE EVENTS:
Time Frame: Date treatment consent signed to date off study, approximately 22 mos./2 days; 13 mos./20 days; 5 mos./23 days; 17 mos./24 days; 7 mos./5 days; 5 mos./5 days; 5 mos./13 days; and 23 mos./21 days for Dose Level (DL) 1, DL2, DL3, DL3 followed by DL2, DL4, DL4 followed by DL3, DL 4 followed by DL 3 followed by DL2; and DL5 respectively.
Arm/Group | Dose Level (DL) 1: Pazopanib (Paz): 400 mg & ARQ 197: 120 mg | Dose Level 2: Pazopanib: 600 mg & ARQ 197: 120 mg | Dose Level 3: Pazopanib: 600 mg & ARQ 197: 240 mg | DL 3 Followed by DL 2: Pazopanib: 600 mg & ARQ 197: 240 mg Foll/by Pazopanib: 600 mg/ARQ 197:120 mg | Dose Level 4: Pazopanib: 800 mg & ARQ 197: 240 mg | DL 4 Followed by DL 3: Pazopanib: 800 mg & ARQ 197: 240 mg Foll/by Pazopanib: 600 mg/ARQ 197: 240 mg | DL4 Foll/by DL3 Foll/by DL2 Paz800mg/ARQ240mg Foll/by Paz600 mg/ARQ240mg Foll/by Paz600 mg/ARQ120 mg | Dose Level 5: Pazopanib: 800 mg & ARQ 197: 360 mg
All-Cause Mortality (participants affected / at risk) | 1/3 | 0/3 | 1/2 | 0/1 | 0/4 | 0/1 | 0/1 | 0/16
Serious Adverse Events (participants affected / at risk) | 1/3 | 2/3 | 1/2 | 0/1 | 1/4 | 0/1 | 0/1 | 6/16
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3 | 2/2 | 1/1 | 4/4 | 1/1 | 1/1 | 16/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dose Level (DL) 1: Pazopanib (Paz): 400 mg & ARQ 197: 120 mg (N=3) | Dose Level 2: Pazopanib: 600 mg & ARQ 197: 120 mg (N=3) | Dose Level 3: Pazopanib: 600 mg & ARQ 197: 240 mg (N=2) | DL 3 Followed by DL 2: Pazopanib: 600 mg & ARQ 197: 240 mg Foll/by Pazopanib: 600 mg/ARQ 197:120 mg (N=1) | Dose Level 4: Pazopanib: 800 mg & ARQ 197: 240 mg (N=4) | DL 4 Followed by DL 3: Pazopanib: 800 mg & ARQ 197: 240 mg Foll/by Pazopanib: 600 mg/ARQ 197: 240 mg (N=1) | DL4 Foll/by DL3 Foll/by DL2 Paz800mg/ARQ240mg Foll/by Paz600 mg/ARQ240mg Foll/by Paz600 mg/ARQ120 mg (N=1) | Dose Level 5: Pazopanib: 800 mg & ARQ 197: 360 mg (N=16)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Alkaline phosphatase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Anorexia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ascites (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Confusion (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Enterocolitis infectious (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Febrile neutropenia (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Fever (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Malaise (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (3)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, death (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, progressive disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pericardial effusion (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary tract obstruction (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (2)
White blood cell decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dose Level (DL) 1: Pazopanib (Paz): 400 mg & ARQ 197: 120 mg (N=3) | Dose Level 2: Pazopanib: 600 mg & ARQ 197: 120 mg (N=3) | Dose Level 3: Pazopanib: 600 mg & ARQ 197: 240 mg (N=2) | DL 3 Followed by DL 2: Pazopanib: 600 mg & ARQ 197: 240 mg Foll/by Pazopanib: 600 mg/ARQ 197:120 mg (N=1) | Dose Level 4: Pazopanib: 800 mg & ARQ 197: 240 mg (N=4) | DL 4 Followed by DL 3: Pazopanib: 800 mg & ARQ 197: 240 mg Foll/by Pazopanib: 600 mg/ARQ 197: 240 mg (N=1) | DL4 Foll/by DL3 Foll/by DL2 Paz800mg/ARQ240mg Foll/by Paz600 mg/ARQ240mg Foll/by Paz600 mg/ARQ120 mg (N=1) | Dose Level 5: Pazopanib: 800 mg & ARQ 197: 360 mg (N=16)
Abdominal pain (Gastrointestinal disorders) | 1 (6) | 1 (3) | 0 (0) | 1 (4) | 0 (0) | 0 (0) | 0 (0) | 4 (5)
Activated partial thromboplastin time prolonged (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Alanine aminotransferase increased (Investigations) | 1 (1) | 1 (2) | 1 (1) | 1 (1) | 2 (3) | 1 (4) | 1 (1) | 2 (4)
Alkaline phosphatase increased (Investigations) | 0 (0) | 2 (3) | 2 (2) | 0 (0) | 2 (3) | 1 (3) | 0 (0) | 6 (10)
Allergic reaction (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
Anal hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 2 (5) | 1 (3) | 1 (1) | 7 (11)
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Metabolism and nutrition disorders) | 1 (2) | 2 (3) | 2 (3) | 1 (1) | 2 (5) | 1 (4) | 1 (2) | 6 (8)
Atrial fibrillation (Cardiac disorders) | 1 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Bloating (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Blood bilirubin increased (Investigations) | 1 (2) | 2 (3) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 6 (9)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Bronchial obstruction (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bruising (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cardiac disorders - Other, non cardiac chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chills (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 3 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (2)
Creatinine increased (Investigations) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (4)
Dehydration (Metabolism and nutrition disorders) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4)
Diarrhea (Gastrointestinal disorders) | 3 (9) | 2 (9) | 1 (3) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 6 (10)
Dizziness (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 3 (3)
Dysgeusia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Edema face (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Edema limbs (General disorders) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Electrocardiogram QT corrected interval prolonged (Cardiac disorders) | 1 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Eye disorders - Other, diplopia (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eye disorders - Other, eye irritation (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 2 (2) | 1 (3) | 1 (1) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 4 (6)
Fever (General disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (4)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Flatulence (Gastrointestinal disorders) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Floaters (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Flu like symptoms (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Flushing (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 7 (7)
Hearing impaired (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Hemoglobinuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Hemorrhoidal hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Hypercalcemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 2 (3)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3)
Hypermagnesemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Hypernatremia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 3 (85) | 3 (45) | 2 (56) | 1 (11) | 3 (87) | 0 (0) | 1 (49) | 13 (188)
Hypoalbuminemia (Metabolism and nutrition disorders) | 2 (4) | 2 (4) | 1 (1) | 0 (0) | 2 (3) | 1 (2) | 0 (0) | 12 (28)
Hypocalcemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 2 (2)
Hypoglycemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypomagnesemia (Metabolism and nutrition disorders) | 1 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 7 (8)
Hypophosphatemia (Metabolism and nutrition disorders) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 5 (6)
Hypothyroidism (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Irregular menstruation (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lip infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lymphocyte count decreased (Investigations) | 3 (16) | 2 (3) | 1 (4) | 0 (0) | 3 (5) | 1 (3) | 1 (8) | 9 (22)
Malaise (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Mucositis oral (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Nausea (Gastrointestinal disorders) | 1 (3) | 2 (3) | 1 (2) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 5 (5)
Neutrophil count decreased (Investigations) | 2 (4) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (4) | 1 (8) | 7 (12)
Non-cardiac chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Otitis externa (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pain of skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Paresthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pelvic pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Platelet count decreased (Investigations) | 1 (1) | 2 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (3) | 3 (6)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Proteinuria (Renal and urinary disorders) | 1 (5) | 2 (3) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 4 (4)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rash acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rectal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Renal and urinary disorders - Other, Dysuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Respiratory, thoracic and mediastinal disorders - Other, chest congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Scalp pain (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sinus bradycardia (Cardiac disorders) | 2 (4) | 1 (1) | 1 (2) | 1 (4) | 4 (11) | 1 (2) | 0 (0) | 11 (18)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin and subcutaneous tissue disorders - Other, Graying of hair (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 2 (2)
Skin and subcutaneous tissue disorders - Other, hair hypopigmentation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin and subcutaneous tissue disorders - Other, skin/hair graying (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin and subcutaneous tissue disorders - Other, whitening of hair (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin and subcutaneous tissue disorders - Other, hypo pigmented of facial hair (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Somnolence (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Stomach pain (Gastrointestinal disorders) | 1 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Trismus (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (6) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (4)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ventricular arrhythmia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (2) | 3 (3) | 0 (0) | 1 (3) | 1 (1) | 1 (2) | 0 (0) | 4 (7)
Weight gain (Investigations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Weight loss (Investigations) | 0 (0) | 1 (3) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
White blood cell decreased (Investigations) | 3 (12) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 1 (4) | 1 (6) | 8 (21)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2017-10-16): https://cdn.clinicaltrials.gov/large-docs/22/NCT01468922/Prot_SAP_000.pdf
  • Informed Consent Form (2015-04-01): https://cdn.clinicaltrials.gov/large-docs/22/NCT01468922/ICF_001.pdf